CLINICAL TRIAL: NCT03086551
Title: Modulating Interaction of Motor Learning Networks in Rehabilitation of Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sean Meehan, Assistant Professor, University of Waterloo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R03NS096484-01 (NIH)
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Stroke, Chronic; Stroke, Middle Cerebral Artery With Infarction
Keywords: Transcranial Magnetic Stimulation; Motor Impairment; Rehabilitation; Motor Learning
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental (Experimental): Application of active continuous theta burst stimulation over dorsolateral prefrontal cortex prior to upper limb motor practice.
  Interventions: Device: Active continuous theta burst stimulation (cTBS); Behavioral: Motor Practice
- Control (Placebo Comparator): Application of sham continuous theta burst stimulation over dorsolateral prefrontal cortex prior to upper limb motor practice.
  Interventions: Device: Placebo (Sham) continuous theta burst stimulation; Behavioral: Motor Practice

INTERVENTIONS:
Device: Active continuous theta burst stimulation (cTBS) — Active cTBS over dorsolateral prefrontal cortex that has an effect upon dorsolateral prefrontal cortex brain activity.
  Arms: Experimental
Device: Placebo (Sham) continuous theta burst stimulation — Sham stimulation over dorsolateral prefrontal cortex that looks and sounds like active cTBS but does not have any effect upon dorsolateral prefrontal cortex brain activity.
  Arms: Control
Behavioral: Motor Practice — Upper limb reaching task to be practiced. Practice will be paired with Active/Sham stimulation. Twenty trials will occur before Active/Sham stimulation. 40 trials will be practiced after Active/Sham stimulation.

SUMMARY:
This study uses a form on non-invasive brain stimulation called transcranial magnetic stimulation to understand 1) understand how the brain learns post-stroke and 2) assess non-invasive brain stimulation as an addition to current stroke rehabilitation approaches. In two study arms the investigators will compare the effect of active transcranial magnetic stimulation paired with motor practice with placebo (or sham) transcranial magnetic stimulation paired with the same motor practice.

DETAILED DESCRIPTION:
Stroke is the leading cause of permanent disability in the United States. In the absence of treatments to restore the lost tissue, clinical scientists have focused upon repetitive forced used of the paretic limb to promote neural reorganization in preserved tissue and reduce disability. However, forced use interventions are time intensive and the extent of functional recovery is variable. One potential contributor to this variability is the potential trade-off between compensatory cognitive motor control strategies and the extent of procedural learning that can occur. Compensatory strategies adopted by patients may produce quick short-term increases in performance but retard slower sustained improvements by interfering with development of procedural learning. Consistent with this hypothesis, the investigators' previous work documents an increased reliance upon dorsolateral prefrontal cortex during performance of learned skills post-stoke. However, the investigators' previous work also demonstrates that the effect of increased activity in dorsolateral prefrontal cortex may limit reorganization in important areas involved in the consolidation of practice thereby limiting functional recovery post-stroke.

Transcranial magnetic stimulation offers a unique opportunity to investigate the relationship between dorsolateral prefrontal cortex activity and consolidation of motor practice/rehabilitaion post-stroke. Here the investigators' objective is to determine whether suppression of the contralesional dorsolateral prefrontal cortex, with continuous theta burst transcranial magnetic brain stimulation (cTBS), a form of transcranial magnetic stimulation, prior to motor practice enhances brain reorganization in critical areas and leads to greater sustained improvements in motor ability over time.

The proposed work will enhance the understanding of motor learning post-stroke and provide preliminary evidence for the benefits of dorsolateral prefrontal cTBS as an adjunct to current rehabilitation interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50-75 years
2. movement-related deficit associated with first time middle cerebral artery stroke
3. greater than 6-months post-stroke
4. Fugl-Meyer score between 15 and 60
5. ability to elicit a motor evoked potential from the ipsilesional cortex

Exclusion Criteria:

1. a score <27 on the Mini-Mental Status Exam
2. a score of <123 on the Mattis Dementia Rating Scale
3. a score of <13 on the Frenchay Aphasia Screen
4. a history of seizure/epilepsy, head trauma, major psychiatric diagnosis, neurodegenerative disorder or substance abuse
5. a history of congestive heart failure
6. systolic blood pressure above 120 mmHg and/or diastolic pressure above 80 mmHg
7. the taking of any GABAergic, NMDA-receptor antagonist or other drug known to influence the neural receptors that facilitate neural plasticity
8. an infarct resulting from ischemic stroke of anterior or posterior cerebral artery OR an infarct that encroaches within 2cm of the site of cTBS stimulation
9. absence of an MEP in response to single pulse transcranial magnetic stimulation over ipsilesional M1 and 10) any other contraindication to TMS or MRI.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean K Meehan, PhD, Principal Investigator — Sch. of Kinesiology, Univ. of Michigan
Locations (1):
- Human Sensorimotor Laboratory, School of Kinesiology, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meehan SK, Randhawa B, Wessel B, Boyd LA. Implicit sequence-specific motor learning after subcortical stroke is associated with increased prefrontal brain activations: an fMRI study. Hum Brain Mapp. 2011 Feb;32(2):290-303. doi: 10.1002/hbm.21019. PMID 20725908
- [Background] Meehan SK, Dao E, Linsdell MA, Boyd LA. Continuous theta burst stimulation over the contralesional sensory and motor cortex enhances motor learning post-stroke. Neurosci Lett. 2011 Aug 1;500(1):26-30. doi: 10.1016/j.neulet.2011.05.237. Epub 2011 Jun 12. PMID 21683125
- [Background] Brodie SM, Meehan S, Borich MR, Boyd LA. 5 Hz repetitive transcranial magnetic stimulation over the ipsilesional sensory cortex enhances motor learning after stroke. Front Hum Neurosci. 2014 Mar 21;8:143. doi: 10.3389/fnhum.2014.00143. eCollection 2014. PMID 24711790
- See also: Primary Investigator's Profile Page — https://uwaterloo.ca/kinesiology/people-profiles/sean-meehan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted through mailings to individuals identified as having been admitted to the University of Michigan Health System in the past 5 years (from 01/01/2012 to 01/27/2017) for treatment of middle cerebral artery stroke. Mailings were sent to those individuals with zip codes in the state of Michigan and northwest Ohio.
Pre-assignment Details: Enrolled participants were excluded prior to randomization for: known contraindication to the transcranial magnetic stimulation intervention (n=1) and a broken foot, not study related, between enrollment and randomization (n=1).
Groups:
- Active+Motor Practice, Then Sham+Motor Practice: Participants first completed four sessions in which motor practice was preceded by ACTIVE continuous theta burst stimulation (cTBS) over dorsolateral prefrontal cortex. After a three-week washout period participants then completed four sessions in which motor practice was preceded by SHAM continuous theta burst stimulation over dorsolateral prefrontal cortex.
- Sham+Motor Practice, Then Active+Motor Practice: Participants first completed four sessions in which motor practice was preceded by SHAM continuous theta burst stimulation (cTBS) over dorsolateral prefrontal cortex. After a three-week washout period participants then completed four sessions in which motor practice was preceded by ACTIVE continuous theta burst stimulation over dorsolateral prefrontal cortex.
Period: First Intervention
Arm/Group | Active+Motor Practice, Then Sham+Motor Practice | Sham+Motor Practice, Then Active+Motor Practice
Started | 5 | 5
Completed | 4 | 4
Not Completed | 1 | 1
Not completed — Failure to meet inclusion criterion | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Washout
Arm/Group | Active+Motor Practice, Then Sham+Motor Practice | Sham+Motor Practice, Then Active+Motor Practice
Started | 4 | 4
Completed | 1 | 1
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Period: Second Intervention
Arm/Group | Active+Motor Practice, Then Sham+Motor Practice | Sham+Motor Practice, Then Active+Motor Practice
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis was completed on all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active+Motor Practice, Then Sham+Motor Practice | Sham+Motor Practice, Then Active+Motor Practice | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10) | 59 (10) | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Fugl-Meyer Assessment of Motor Recovery After Stroke (Upper Limb) [Mean (Standard Deviation); unit: units on a scale] — The Fugl-Meyer Assessment of Motor Recovery After Stroke (Upper Limb) scale is a stroke-specific scale designed to assess motor functioning in patients with post-stroke hemiplegia. The upper limb scale ranges between 0 (severe functional impairment) to 66 (minimal functional impairment)
  units on a scale | 50 (17) | 48 (24) | 49 (20)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment is a questionnaire used to assess cognitive impairment. The test has a scale that ranges between 0 (severe cognitive impairment) and 30 (typical cognitive function).
  units on a scale | 28 (2) | 24 (3) | 26 (3)
Mini-Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination is used in clinical and research settings to measure cognitive impairment. The scale ranges from 0 (severe cognitive impairment) to 30 (no cognitive impairment).
  units on a scale | 30 (1) | 27 (3) | 29 (2)
Trail Making Test A [Mean (Standard Deviation); unit: seconds] — Trail Making Test A is a timed test that assesses cognitive processing speed. The participant is required to draw lines to connect a sequence of twenty-five consecutively numbered targets (1, 2, 3, etc.) on a sheet of paper. If the subject makes an error, the test administrator corrects them before the subject moves on to the next numbered target.
  seconds | 29.6 (6.9) | 31.1 (13.3) | 30.3 (9.5)
Trail Making Test B [Mean (Standard Deviation); unit: seconds] — Trail Making Test B is a timed test used to assess executive functioning. The participant is required to draw lines to connect a series of targets labelled by either a number or letter in sequential order. When connecting the targets the participant alternates between numbers and letters (1, A, 2, B, etc.). If the subject makes an error, the test administrator corrects them before the participant moves on to the next dot.
  seconds | 29.6 (33.1) | 89.7 (26.2) | 75.3 (31.1)
Stroke Affected Hemisphere [Count of Participants; unit: Participants] — Count of stroke affected hemisphere
  Participants
    Left Hemisphere | 2 | 4 | 6
    Right Hemisphere | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sequential Response Time to Post-Intervention
Description: Aggregate time to complete movements between a six sequential targets presented on a computer touch screen in front of the participant. The mean of ten sequences was calculated prior to any practice and at a delayed retention test (e.g. no warm up or preceding practice) post-intervention. Change between the baseline average and post-intervention average was also calculated by subtracting post-intervention score from pre-intervention score. Positive numbers represent improvement in ability.
Time Frame: Baseline and post-intervention
Population: All participants who completed at least one arm of the study
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Active+Motor Practice: Participants who received motor practice preceded by ACTIVE continuous theta burst stimulation (cTBS) over dorsolateral prefrontal cortex in either the first three weeks or last three weeks of the study.
- Sham+Motor Practice: Participants who received motor practice preceded by SHAM continuous theta burst stimulation (cTBS) over dorsolateral prefrontal cortex in either the first three weeks or last three weeks of the study.
Arm/Group | Active+Motor Practice | Sham+Motor Practice
Number analyzed (Participants) | 5 | 5
seconds
  Time to Complete Sequence (Baseline) | 8.68 (2.06) | 8.84 (1.47)
  Time to Complete Sequence (Delayed Retention) | 8.32 (1.55) | 7.96 (1.04)
  Change in Time (Pre to Post) | 0.37 (0.65) | 0.88 (0.63)
Statistical Analysis 1: Comparison: Active+Motor Practice vs Sham+Motor Practice; Magnitude of change in sequence completion time from pre-baseline to post-intervention for the Active arm. Cohen's d was calculated as a measure of effect size; Test type: Other; Effect Size - Cohen's d = 0.20 — Cohen's d was calculated as time to complete the sequence at the pre-baseline assessment minus the time it took to complete the sequence at the post-intervention assessment. The denominator reflected pooled variance
Statistical Analysis 2: Comparison: Active+Motor Practice vs Sham+Motor Practice; Magnitude of change in sequence completion time from pre-baseline to post-intervention for the Sham arm. Cohen's d was calculated as a measure of effect size; Test type: Other; Effect Size - Cohen's d = 0.69 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Active+Motor Practice vs Sham+Motor Practice; Test type: Other — Cohen's d effect size was calculated to compare the magnitude of change in time to complete the movement sequence from pre-baseline to post-intervention across the Active and Sham arms; Effect Size - Cohen's d = -0.80 — Cohen's d was calculated as the change from pre- to post-intervention for the Active arm minus change from pre- to post-intervention for the Sham arm. The denominator reflected pooled variance

2. Secondary Outcome: Change From Baseline in Time to Complete the Jebsen-Taylor Hand Function Test
Description: The Jebsen-Taylor Hand Function Test is comprised of a series of unimanual tasks required for activities of daily living. Time to complete the Jebsen-Taylor Hand Function Test was assessed at baseline and post-intervention by taking the aggregate time to complete each activity. Change in time to complete the Jebsen-Taylor Hand Function Test between the baseline and post-intervention tests was derived by subtracting post-intervention score from baseline score. Positive scores indicate improvement in functional motor ability.
Time Frame: Baseline and post-intervention
Population: All participants who completed at least one arm of the study
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active+Motor Practice | Sham+Motor Practice
Number analyzed (Participants) | 5 | 5
seconds
  Pre Time to Complete (Stroke Affected Limb) | 95.68 (51.71) | 86.07 (17.78)
  Post Time to Complete (Stroke Affected Limb) | 100.05 (60.47) | 76.27 (20.97)
  Change Pre to Post (Stroke Affected Limb) | -4.38 (8.95) | 9.80 (6.14)
  Pre Time to Complete (Non-Stroke Affected Limb) | 55.75 (11.22) | 66.67 (20.87)
  Post Time to Complete (Non-Stroke Affected Limb) | 51.97 (8.25) | 64.95 (24.07)
  Change Pre to Post (Non-Stroke Affected Limb) | 3.78 (5.33) | 1.72 (5.40)
Statistical Analysis 1: Comparison: Active+Motor Practice vs Sham+Motor Practice; The magnitude of transfer of the task specific practice to functional activities of daily live for the stroke affected limb was assessed by calculating the magnitude of change (Cohen's d) in time to complete the activities of the Jebsen-Taylor Hand Function Test from pre-baseline to post-intervention in the Active arm; Test type: Other; Effect Size - Cohen's d = -0.08 — Cohen's d was calculated as aggregate time to complete all elements at the pre-baseline assessment minus the aggregate time it took to complete all elements at the post-intervention assessment. The denominator reflected pooled variance
Statistical Analysis 2: Comparison: Active+Motor Practice vs Sham+Motor Practice; The magnitude of transfer of the task specific practice to functional activities of daily live for the stroke affected limb was assessed by calculating the magnitude of change (Cohen's d) in time to complete the activities of the Jebsen-Taylor Hand Function Test from pre-baseline to post-intervention in the Sham arm; Test type: Other; Effect Size - Cohen's d = 0.50 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Active+Motor Practice vs Sham+Motor Practice; Comparison across study arm of the magnitude of improvement in aggregate time to complete all elements of the Jebsen-Taylor Hand Function Test for the stroke affected limb. Cohen's d was calculated as a measure of effect size; Test type: Other; Effect Size - Cohen's d = -1.84 — Cohen's d was calculated as the change from pre- to post-intervention for the Active arm minus the change from pre- to post-intervention for the Sham arm. The denominator reflected pooled variance
Statistical Analysis 4: Comparison: Active+Motor Practice vs Sham+Motor Practice; The magnitude of transfer of the task specific practice to functional activities of daily live for the non-stroke affected limb was assessed by calculating the magnitude of change (Cohen's d) in time to complete the activities of the Jebsen-Taylor Hand Function Test from pre-baseline to post-intervention in the Active arm; Test type: Other; Effect Size - Cohen's d = 0.38 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Active+Motor Practice vs Sham+Motor Practice; The magnitude of transfer of the task specific practice to functional activities of daily live for the non-stroke affected limb was assessed by calculating the magnitude of change (Cohen's d) in time to complete the activities of the Jebsen-Taylor Hand Function Test from pre-baseline to post-intervention in the Sham arm; Test type: Other; Effect Size - Cohen's d = 0.08 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Active+Motor Practice vs Sham+Motor Practice; Comparison across study arm of the magnitude of improvement in aggregate time to complete all elements of the Jebsen-Taylor Hand Function Test for the non-stroke affected limb. Cohen's d was calculated as a measure of effect size; Test type: Other; Effect Size - Cohen's d = 0.38 — [estimate comment as in outcome 2, analysis 3]

3. Secondary Outcome: Change in Sequential Response Time Immediately Follow an Individual Bout of Non-invasive Brain Stimulation (e.g. Within Session)
Description: Aggregate time to complete movements between a six sequential targets presented on a computer touch screen in front of the participant. The mean of ten sequences was calculated prior to application of Active+Motor Practice or Sham+Motor Practice for each intervention session and the first ten sequences of practice immediately following the specific form of non-invasive brain stimulation within each session. Change within a session was calculated by subtracting the post-stimulation score from the pre-stimulation score within a session. Positive values represent improved ability.
Time Frame: Within session baseline to ~8 minutes post-application of non-invasive stimulation within the same session
Population: All participants who completed at least one arm of the study
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active+Motor Practice | Sham+Motor Practice
Number analyzed (Participants) | 5 | 5
seconds
  Session 1 | 0.41 (0.70) | 0.89 (0.36)
  Session 2 | 0.72 (1.97) | 0.80 (1.86)
  Session 3 | -0.20 (0.60) | 0.22 (0.62)
  Session 4 | 0.35 (0.46) | 0.23 (0.39)
Statistical Analysis 1: Comparison: Active+Motor Practice vs Sham+Motor Practice; The immediate effect of continuous theta burst stimulation over dorsolateral prefrontal cortex prior to practice was assessed by determining the magnitude of the effect of Active stimulation from pre-intervention to immediately post-intervention in Session 1 of the intervention. Cohen's d was used to derive effect size. The Sham stimulation change was used as the control; Test type: Other; Effect Size - Cohen's d = -0.86 — Cohen's d was calculated as the change from pre- to immediately post-stimulation (within the same session) for the Active arm minus the change from pre- to immediately post-stimulation for the Sham arm. The denominator reflected pooled variance
Statistical Analysis 2: Comparison: Active+Motor Practice vs Sham+Motor Practice; The immediate effect of continuous theta burst stimulation over dorsolateral prefrontal cortex prior to practice was assessed by determining the magnitude of the effect of Active stimulation from pre-intervention to immediately post-intervention in Session 2 of the intervention. Cohen's d was used to derive effect size. The Sham stimulation change was used as the control; Test type: Other; Effect Size - Cohen's d = -0.04 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Active+Motor Practice vs Sham+Motor Practice; The immediate effect of continuous theta burst stimulation over dorsolateral prefrontal cortex prior to practice was assessed by determining the magnitude of the effect of Active stimulation from pre-intervention to immediately post-intervention in Session 3 of the intervention. Cohen's d was used to derive effect size. The Sham stimulation change was used as the control; Test type: Other; Effect Size - Cohen's d = -0.69 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Active+Motor Practice vs Sham+Motor Practice; The immediate effect of continuous theta burst stimulation over dorsolateral prefrontal cortex prior to practice was assessed by determining the magnitude of the effect of Active stimulation from pre-intervention to immediately post-intervention in Session 4 of the intervention. Cohen's d was used to derive effect size. The Sham stimulation change was used as the control; Test type: Other; Effect Size - Cohen's d = 0.28 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Motor Evoked Potential Amplitude (in Microvolts) at Pre-baseline and Post-Intervention
Description: Motor evoked potential amplitude evoked by transcranial magnetic brain stimulation was recorded using electromyography over the first dorsal interosseous muscle of the stroke-affected hand. The means of ten trials at 120% (linear part of recruitment curve) and ten trials at 150% (recruitment curve plateau) of resting motor threshold were calculated and expressed in microvolts.
Time Frame: Baseline and post-intervention
Population: All participants who completed at least one arm of the study
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Active+Motor Practice | Sham+Motor Practice
Number analyzed (Participants) | 5 | 5
microvolts
  MEP Amplitude Pre (120% of RMT) | 1558 (1020) | 971 (709)
  MEP Amplitude Post (120% of RMT) | 1216 (1161) | 511 (279)
  MEP Amplitude Pre (150% of RMT) | 2750 (2172) | 1977 (218)
  MEP Amplitude Post (150% of RMT) | 2008 (2062) | 2495 (609)
Statistical Analysis 1: Comparison: Active+Motor Practice vs Sham+Motor Practice; Comparison of first dorsal interosseous motor evoked potential (MEP) amplitude elicited from the ipsilesional motor cortex pre-baseline to post-intervention for the Active arm when transcranial magnetic stimulator intensity was set to 120% of resting motor threshold. Estimate of effect size was derived using Cohen's d; Test type: Other; Effect Size - Cohen's d = -0.31 — Cohen's d was calculated as the amplitude of the motor evoked potential at the post-intervention assessment minus the amplitude of the motor evoked potential at the pre-baseline assessment. The denominator reflected pooled variance
Statistical Analysis 2: Comparison: Active+Motor Practice vs Sham+Motor Practice; Comparison of first dorsal interosseous motor evoked potential (MEP) amplitude elicited from the ipsilesional motor cortex pre-baseline to post-intervention for the Sham arm when transcranial magnetic stimulator intensity was set to 120% of resting motor threshold. Estimate of effect size was derived using Cohen's d; Test type: Other; Effect Size - Cohen's d = -0.85 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Active+Motor Practice vs Sham+Motor Practice; Comparison of the first dorsal interosseous motor evoked potential (MEP) amplitude elicited from the ipsilesional motor cortex pre-baseline to post-intervention for the Active arm when transcranial magnetic stimulator intensity was set to 150% of resting motor threshold. Estimate of effect size was derived using Cohen's d; Test type: Other; Effect Size - Cohen's d = -0.35 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Active+Motor Practice vs Sham+Motor Practice; Comparison of the first dorsal interosseous motor evoked potential (MEP) amplitude elicited from the ipsilesional motor cortex pre-baseline to post-intervention for the Sham arm when transcranial magnetic stimulator intensity was set to 150% of resting motor threshold. Estimate of effect size was derived using Cohen's d; Test type: Other; Effect Size - Cohen's d = 1.13 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Cortical Excitability Post-Intervention
Description: Motor evoked potential amplitude evoked by transcranial magnetic brain stimulation was recorded using electromyography over the first dorsal interosseous muscle of the stroke-affected hand. The means of ten trials at 120% (linear part of recruitment curve) and ten trials at 150% (recruitment curve plateau) of resting motor threshold were calculated and expressed in microvolts. Change in motor evoked potential amplitude elicited by transcranial magnetic stimulation intensities of 120% (linear part of recruitment curve) and ten trials at 150% (recruitment curve plateau) of resting motor threshold. Values are expressed percent change relative to pre-baseline values. Positive numbers represent an increase motor evoked potential from pre-baseline to post-intervention.
Time Frame: Baseline and post-intervention
Population: All participants who completed at least one arm of the study
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Active+Motor Practice | Sham+Motor Practice
Number analyzed (Participants) | 5 | 5
percentage change
  % change in MEP (120% RMT) | -26 (35) | -19 (58)
  % change in MEP (150% RMT) | -17 (37) | 25 (17)
Statistical Analysis 1: Comparison: Active+Motor Practice vs Sham+Motor Practice; Comparison of the first dorsal interosseous motor evoked potential (MEP) amplitude elicited from the ipsilesional motor cortex pre-baseline to post-intervention across the Active and Sham arms when transcranial magnetic stimulator intensity was set to 120% of resting motor threshold. Comparison quantified as effect size using Cohen's d; Test type: Other; Effect Size - Cohen's d = -0.15 — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 2: Comparison: Active+Motor Practice vs Sham+Motor Practice; Comparison of the first dorsal interosseous motor evoked potential (MEP) amplitude elicited from the ipsilesional motor cortex pre-baseline to post-intervention across the Active and Sham arms when transcranial magnetic stimulator intensity was set to 150% of resting motor threshold. Comparison quantified as effect size using Cohen's d; Test type: Other; Effect Size - Cohen's d = -1.46 — [estimate comment as in outcome 2, analysis 3]

ADVERSE EVENTS:
Time Frame: Duration of study (9 weeks)
Description: The total numbers reported reflect all participants who completed at least one session of the intervention.
Arm/Group | Active+Motor Practice | Sham+Motor Practice
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT03086551/Prot_SAP_000.pdf